CLINICAL TRIAL: NCT03962374
Title: The Comparison of the Success Rate of the Endotracheal Intubation Between the Stylet and the Frova With Acute Angled Videolaryngoscope
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4-2019-0289
Record Dates: First submitted 2019-05-22; First posted 2019-05-24 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-12

CONDITIONS: Anesthesia, General

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Frova (Experimental): Frova will be used to facilitate the endotracheal intubation.
  Interventions: Device: Frova
- Stylet (Active Comparator): Stylet will be used to facilitate the endotracheal intubation.
  Interventions: Device: Stylet

INTERVENTIONS:
Device: Frova — Frova will be used to facilitate the endotracheal intubation. The success rate of first attempt of intubation will be assessed.
  Arms: Frova
Device: Stylet — Stylet will be used to facilitate the endotracheal intubation. The success rate of first attempt of intubation will be assessed.
  Arms: Stylet

SUMMARY:
The purpose of this study is to compare the effect of frova and stylet on the success rate of tracheal intubation when using a video laryngoscope.

ELIGIBILITY:
Inclusion Criteria:

* 1. adult patients aged over 19 years who are undergoing endotracheal intubation for elective surgery.
* 2. Patients who have one of the predictors of difficult intubation such as Mallampati classification 3 or 4, limited the movement of the neck, body mass index less than 35 kg/m2, a distance from the tip of the chin to the thyroid cartilage of less than 6.5 cm, a interincisor distance less than 3.5 cm, inability to protrude of lower incisors over the upper incisors, or a diagnosis of obstructive sleep apnea.

Exclusion Criteria:

* 1. Patients receiving emergency surgery
* 2. Pregnant women
* 3. Patients scheduled for oral surgery such as tonsillectomy, vocal cord surgery
* 4. Patients who have a history of ankylosing spondylitis or have a large tumor of 4 cm or more on the tongue and need an awake intubation
* 5. Patients who are at risk of vomiting due to not fasting time

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Estimated)
Dates: Start 2022-06-21 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Success rate of first attempt of endotracheal intubation | for 10 minutes during anesthetic induction
  The endotracheal intubation will be attempted using stylet or frova according to the randomized group. The success or failure of the attempt will be recorded.

SECONDARY OUTCOMES:
time for endotracheal intubation | for 10 minutes during anesthetic induction
  Time will be measured from when the blades of the videolaryngoscope pass through the patient's mouth until the end-tidal CO2 is detected.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institute, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No